CLINICAL TRIAL: NCT02116608
Title: Treatment of Tracheostomy Granulomas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2819
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Granuloma; Tracheostomy
MeSH Terms: conditions — Granuloma | interventions — Povidone-Iodine; Silver Nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Betadine (Active Comparator): Apply locally as needed.
  Interventions: Drug: Betadine
- Group 2: Silver Nitrate (Active Comparator): Arzol Silver Nitrate Applicators may be applied directly to mucous membranes and other moist surfaces. In the case of dry skin, the applicator tip should be dipped in water immediately before use. Apply carefully to the area to be treated.
  Interventions: Drug: Silver Nitrate
- Group 3: Hydrocortisone Butyrate Cream, 1.0% (Active Comparator): Hydrocortisone butyrate cream, 1.0% should be applied to the affected area as a thin film two or three times daily depending on the severity of the condition.
  Interventions: Drug: Hydrocortisone Butyrate Cream, 1.0%

INTERVENTIONS:
Drug: Betadine — Apply locally as needed.
  Arms: Group 1: Betadine
Drug: Silver Nitrate — Arzol Silver Nitrate Applicators may be applied directly to mucous membranes and other moist surfaces. In the case of dry skin, the applicator tip should be dipped in water immediately before use. Apply carefully to the area to be treated.
  Arms: Group 2: Silver Nitrate
Drug: Hydrocortisone Butyrate Cream, 1.0% — Hydrocortisone butyrate cream, 1.0% should be applied to the affected area as a thin film two or three times daily depending on the severity of the condition.
  Arms: Group 3: Hydrocortisone Butyrate Cream, 1.0%

SUMMARY:
This study plans to learn more about the different ways used to treat tracheostomy granulomas. Investigators want to see which standard of care method (steroid application, silver nitrate, or betadine) is more successful in treating tracheostomy granulomas.

DETAILED DESCRIPTION:
Upon joining the study patients will be assigned to one of the three treatment groups (steroid application, silver nitrate, and betadine). These three treatments are standard of care and patients would have been treated with one of them anyway. Patients will be followed for an observation period of six weeks with follow-up appointments, per standard of care, every two weeks (+/- 3 days) in order for a physician to evaluate if the treatment method is working. If during a follow-up visit, the physician determines the treatment method is not working, the follow-up period will end and participation in the study will be complete. In addition, if a patient is given a different form of treatment during the observation period, such as in the emergency department or through their primary care physician, the follow-up period will end and participation in the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Children's Hospital Colorado inpatient or outpatient
* 31 days to 17 years (inclusive)
* Needs treatment for a tracheostomy granuloma

Exclusion Criteria:

* Tracheostomy granuloma has been treated in the last two weeks

Ages: 31 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Prager, MD, Principal Investigator — 1. University of Colorado School of Medicine, Department of Otolaryngology 2. Children's Hospital Colorado, Department of Pediatric Otolaryngology
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaremchuk K. Regular tracheostomy tube changes to prevent formation of granulation tissue. Laryngoscope. 2003 Jan;113(1):1-10. doi: 10.1097/00005537-200301000-00001. PMID 12514373
- [Background] Chen C, Bent JP, Parikh SR. Powered debridement of suprastomal granulation tissue to facilitate pediatric tracheotomy decannulation. Int J Pediatr Otorhinolaryngol. 2011 Dec;75(12):1558-61. doi: 10.1016/j.ijporl.2011.09.007. Epub 2011 Oct 11. PMID 21996151
- [Background] Al-Samri M, Mitchell I, Drummond DS, Bjornson C. Tracheostomy in children: a population-based experience over 17 years. Pediatr Pulmonol. 2010 May;45(5):487-93. doi: 10.1002/ppul.21206. PMID 20425857
- [Background] McShane DB, Bellet JS. Treatment of hypergranulation tissue with high potency topical corticosteroids in children. Pediatr Dermatol. 2012 Sep-Oct;29(5):675-8. doi: 10.1111/j.1525-1470.2012.01724.x. Epub 2012 May 21. PMID 22612258

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: Hydrocortisone Butyrate Cream, 1.0%: Hydrocortisone butyrate cream, 1.0% should be applied to the affected area as a thin film two or three times daily depending on the severity of the condition.
  Hydrocortisone Butyrate Cream, 1.0%: Hydrocortisone butyrate cream, 1.0% should be applied to the affected area as a thin film two or three times daily depending on the severity of the condition.
- Group 3: Silver Nitrate: Arzol Silver Nitrate Applicators may be applied directly to mucous membranes and other moist surfaces. In the case of dry skin, the applicator tip should be dipped in water immediately before use. Apply carefully to the area to be treated.
  Silver Nitrate: Arzol Silver Nitrate Applicators may be applied directly to mucous membranes and other moist surfaces. In the case of dry skin, the applicator tip should be dipped in water immediately before use. Apply carefully to the area to be treated.
Period: Overall Study
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate
Started | 9 | 9 | 8
Completed | 9 | 7 | 7
Not Completed | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate | Total
Number analyzed (Participants) | 9 | 9 | 8 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 8 | 26
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: days] | 1190.778 [142 to 5534] | 256.333 [128 to 507] | 897.625 [114 to 3771] | 777.115 [114 to 5534]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data was not collected for the 3 participants who did not complete the study.
  Participants
    number analyzed (Participants) | 9 | 7 | 7 | 23
    Hispanic or Latino | 3 | 1 | 1 | 5
    Not Hispanic or Latino | 6 | 6 | 6 | 18
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data was not collected for the 3 participants who did not complete the study.
  Participants
    number analyzed (Participants) | 9 | 7 | 7 | 23
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 2 | 4
    White | 8 | 6 | 3 | 17
    More than one race | 0 | 0 | 2 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Success and Failure Rates for Each Treatment Method
Description: Definition of success: The investigators are defining successful treatment of tracheostomy granulomas as a decrease in the frequency of granulomas over a six week observation period using the assigned treatment or partial or complete resolution of the granuloma. Partial resolution is defined as 25-75% resolution and complete resolution is defined as greater than 75% resolution.
  Definition of failure: The investigators are defining a treatment as a failure if during the six week observation period of using the assigned treatment, there is either no improvement in the resolution or there has been an increase in size or frequency of tracheostomy granulomas.
Time Frame: Over 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate
Number analyzed (Participants) | 9 | 7 | 7
Participants
  Success | 6 | 3 | 5
  Failure | 3 | 4 | 2

2. Primary Outcome: Categorical Improvement (Degree of Improvement)
Description: Categorical success/failure data. the size of the granuloma will be measured and recorded. The percent circumference will also be measured. The approximate percent decrease in the granuloma size will be determined to determine the category subject's change in granuloma:
  i. Complete resolution: >90% improvement (Score = 4) ii. Improvement: 50 - 90% improvement (Score = 3) iii. Minimal improvement: < 50% improvement (Score = 2) iv. No improvement (Score = 1) v. Worsening (Score = 0)
Time Frame: Over 6 Weeks
Population: This outcome measure was initially grouped in error under another outcome measure at registration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate
Number analyzed (Participants) | 9 | 7 | 7
Participants
  Worsening | 0 | 2 | 2
  No improvement | 1 | 1 | 0
  Minimal improvement: < 50% improvement | 2 | 1 | 0
  Improvement: 50-90% improvement | 2 | 0 | 0
  Complete resolution: >90% improvement | 4 | 3 | 5

3. Secondary Outcome: Length of Time Between Administration of the Treatment and the Determination of Treatment Failure, if Applicable
Description: Over the 6 week treatment period, the time from administration of the treatment to the time of treatment failure, if it occurs, will be evaluated and documented.
Time Frame: Over 6 weeks
Population: No data was collected for this outcome measure.
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Group 1: Betadine | Group 2: Hydrocortisone Butyrate Cream, 1.0% | Group 3: Silver Nitrate
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/9 | 1/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Betadine (N=9) | Group 2: Hydrocortisone Butyrate Cream, 1.0% (N=9) | Group 3: Silver Nitrate (N=8)
Death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Viral Respiratory Infection
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02116608/Prot_SAP_000.pdf